CLINICAL TRIAL: NCT07383610
Title: Investigation of Ultrasonographic Predictors of Difficult Intubation and Difficult Mask Ventilation in Adult Patients
Brief Title: Ultrasound Predictors of Difficult Airway in Adults
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Serkan TELLİ, Principal Investigator, Kutahya Health Sciences University
Other Study IDs: 2023/10-19
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Difficult Intubation; Difficult Mask Ventilation; Difficult Airway
Keywords: Airway Ultrasonography; Ultrasound; Difficult Airway Prediction; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Adult patients undergoing surgery under general anesthesia: Adult patients (18-70 years, ASA I-III) scheduled for elective surgery under general anesthesia requiring orotracheal intubation. Preoperative clinical airway assessment and ultrasonographic airway measurements were recorded, and intraoperative intubation and mask ventilation outcomes were evaluated

SUMMARY:
Difficult airway management is a major cause of perioperative complications. Standard bedside airway assessment tests may have limited ability to predict difficult intubation and difficult mask ventilation. This prospective observational study aims to evaluate whether preoperative ultrasound measurements of airway structures (such as skin-to-epiglottis distance, tongue thickness, and pre-epiglottic space) can predict difficult intubation and difficult mask ventilation in adult patients undergoing surgery under general anesthesia.

DETAILED DESCRIPTION:
This prospective observational cohort study was conducted to evaluate the predictive value of preoperative ultrasonographic airway measurements for difficult intubation and difficult mask ventilation in adult patients undergoing elective surgery under general anesthesia. A total of 400 patients aged 18-70 years with ASA physical status I-III were included. Before induction of anesthesia, standard clinical airway assessment tests were recorded, and ultrasound measurements were performed to assess airway-related anatomical structures. Ultrasonographic parameters included skin-to-epiglottis distance, skin-to-thyroid cartilage distance, thyroid cartilage-to-epiglottis distance, pre-epiglottic space depth, tongue thickness, and hyomental distance measurements.

Intraoperatively, mask ventilation and intubation conditions were documented. Difficult intubation was defined as requiring two or more intubation attempts. Difficult mask ventilation was defined as the need for two-handed mask ventilation or inability to ventilate adequately using a face mask. The primary objective was to determine the association between ultrasonographic measurements and difficult intubation

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years

ASA physical status I-III

Elective surgery under general anesthesia requiring orotracheal intubation

Written informed consent

Exclusion Criteria:

* Refusal to participate

Emergency surgery

Pregnancy

Known upper airway pathology or previous airway surgery

Restricted mouth opening (<3 cm)

Cervical spine instability or significant limitation of neck mobility

Morbid obesity (BMI ≥40 kg/m²)

Obstructive upper airway masses (e.g., head and neck tumors)

Prior neck radiotherapy

Clinically relevant neck masses

Major facial/mandibular trauma or craniofacial anomalies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-70 years (ASA I-III) scheduled for elective surgery under general anesthesia requiring orotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Difficult Intubation | During induction of anesthesia (intraoperative)
  Difficult intubation was defined as requiring two or more intubation attempts (≥2 attempts) during induction of general anesthesia.
Number of Participants with Difficult Mask Ventilation | During induction of anesthesia (intraoperative)
  Difficult mask ventilation was defined as the need for two-handed mask ventilation or inability to ventilate adequately using a face mask

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Telli, MD, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional policies and to protect participant privacy and confidentiality.

REFERENCES:
- [Result] 1. Cook TM, MacDougall-Davis SR. Complications and failure of airway management. Br J Anaesth. 2012;109 Suppl 1(suppl 1):i68-i85. 2. Apfelbaum JL, Hagberg CA, Connis RT, Abdelmalak BB, Agarkar M, Dutton RP, et al. 2022 American Society of Anesthesiologists Practice Guidelines for Management of the Difficult Airway. Anesthesiology. 2022;136(1):31-81. 3. Roth D, Pace NL, Lee A, Hovhannisyan K, Warenits AM, Arrich J, et al. Airway physical examination tests for detection of difficult airway management in apparently normal adult patients. Cochrane Database Syst Rev. 2018;5(5):CD008874. 4. Shiga T, Wajima Z, Inoue T, Sakamoto A. Predicting difficult intubation in apparently normal patients: a meta-analysis of bedside screening test performance. Anesthesiology. 2005;103(2):429-37. 5. Detsky ME, Jivraj N, Adhikari NK, Friedrich JO, Pinto R, Simel DL, et al. Will This Patient Be Difficult to Intubate?: The Rational Clinical Examination Systematic Review. JAMA. 2019;321(5):493-503. 6. Singh M, Chin KJ, Chan VW, Wong DT, Prasad GA, Yu E. Use of sonography for airway assessment: an observational study. J Ultrasound Med. 2010;29(1):79-85. 7. Kundra P, Mishra SK, Ramesh A. Ultrasound of the airway. Indian J Anaesth. 2011;55(5):456-62. 8. Marchis IF, Negrut MF, Blebea CM, Crihan M, Alexa AL, Breazu CM. Trends in Preoperative Airway Assessment. Diagnostics (Basel). 2024;14(6). 9. Yao W, Wang B. Can tongue thickness measured by ultrasonography predict difficult tracheal intubation? Br J Anaesth. 2017;118(4):601-9. 10. Daggupati H, Maurya I, Singh RD, Ravishankar M. Development of a scoring system for predicting difficult intubation using ultrasonography. Indian J Anaesth. 2020;64(3):187-92. 11. Sotoodehnia M, Khodayar M, Jalali A, Momeni M, Safaie A, Abdollahi A. Prediction of difficult laryngoscopy / difficult intubation cases using upper airway ultrasound measurements in emergency department: a prospective observational study. BMC Emerg Med. 2023;23(1):78